CLINICAL TRIAL: NCT00110526
Title: Phase I Trial of Adenovirus- Mediated IL-12 Gene Transduction in Patients With Radiorecurrent Prostate Cancer
Brief Title: Gene Therapy for Prostate Cancer That Returns After Radiation Therapy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants met eligibility requirements
Sponsor: Simon Hall (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Simon Hall, MD, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO # 01-0595; A-11425
Record Dates: First submitted 2005-05-10; First posted 2005-05-11 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Prostatic Neoplasms; Neoplasm Recurrence, Local
Keywords: Prostate Cancer; Radiation Therapy; Local recurrence; Gene Therapy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Recurrence, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ad.hIL-12 (Experimental)
  Interventions: Genetic: Ad.hIL-12

INTERVENTIONS:
Genetic: Ad.hIL-12 — Ad.hIL-12 intraprostatic injection IND

SUMMARY:
The purpose of this research study is to test a new treatment for prostate cancer. We have been exploring the use of cytokine (immune stimulating) gene therapy by directly injecting a virus which produces a cytokine called interleukin-12 (IL-12) into the prostate gland to control tumor growth. We propose to explore the use of adenovirus-mediated human interleukin-12 (Ad.hIL-12) in patients with recurrent non-metastatic prostate cancer following radiation therapy in a Phase I trial. Participants will be placed in rising dose groups with the primary endpoint of learning the maximum dose that can safely be given by injection directly into the prostate gland. Toxicity will be determined through physical examination, laboratory values, and blood levels of cytokines. Evidence of an immune response against prostate proteins will also be monitored. If the treatment works, the cancer will shrink or not grow. This will be monitored by prostate specific antigen (PSA) levels in the blood. However, we do not know if this treatment will be effective. If the PSA continues to rise after treatment, participants will be taken off study and offered other treatment. There is no compensation for participation in this research study. There will be no charge for the treatment with gene therapy or the monitoring associated with this research study. Monitoring will occur in a specially designated clinical research center.

DETAILED DESCRIPTION:
Patients with radiorecurrent prostate cancer have few viable treatment options, both in terms of efficacy and morbidity. Local therapies fail even in highly selected patients due to locally advanced disease, microscopic metastases, and a worsening of the biology of cancer cells. Furthermore, attempts at salvage local treatments have the complications of incontinence, impotence and in some cases unremitting penile pain. Pre-clinical studies in a mouse model of prostate cancer have noted the potential benefit of adenovirus-mediated gene therapy to deliver IL-12 in this clinical scenario. This treatment was able to significantly growth suppress the injected tumor to prolong survival and reduce the number of pre-established metastases. The mechanisms underlying this activity involved both innate immunity (neutrophils and natural killer [NK] cells) and acquired immunity ( T cells) and enhanced expression of Fas to further sensitize Fas/Fas ligand (FasL) killing.

This is a Phase I study. Therefore, the primary objective is finding the Maximum Tolerated Dose. Within this realm will be monitoring of pro-inflammatory cytokines. Secondary aspects will involve correlating important mechanisms identified in the pre-clinical model: induction of T cells.

ELIGIBILITY:
Inclusion Criteria:

* A local recurrence of prostate cancer (in or next to gland) following treatment by radiation therapy (either external beam or seed implantation)
* Rising PSA (Prostate Specific Antigen) on at least three occasions separated by two weeks
* Ultrasound guided biopsy to diagnose recurrent disease within the prostate
* No evidence of prostate cancer that has spread on bone scan or Computed Tomography (CT) scan
* No hormone therapy at time of enrollment to the research study

Exclusion Criteria:

* Radical prostatectomy for treatment of prostate cancer
* Detectable spread of prostate cancer on bone or CT scan
* Immunosuppressive medication within two months of the study
* Acute infection (any bacterial, viral, fungal infection requiring specific therapy)
* HIV disease
* Other significant medical or psychiatric conditions which pose high risk for an investigational study

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
maximum cytokine gene therapy level | after 56 weeks, every 6 months up to 15 years
  To study in a Phase I clinical trial the safety of intraprostatic injection of a replication incompetent adenovirus expressing hIL-12 in patients with radiorecurrent prostate cancer

SECONDARY OUTCOMES:
serum pro-inflammatory cytokines levels | up to 15 years
  To assess serum levels of pro-inflammatory cytokines before and after vector injection and will continue every 3 days until normalized
To assess T cell responses pre and post-IL-12 treatment against prostate antigens | Day 7 post vector injection
  Day 7,14,21 and 28 post vector injection
To assess T cell responses pre and post-IL-12 treatment against prostate antigens | Day 14 post vector injection
  Day 7,14,21 and 28 post vector injection
To assess T cell responses pre and post-IL-12 treatment against prostate antigens | Day 21 post vector injection
  Day 7,14,21 and 28 post vector injection
To assess T cell responses pre and post-IL-12 treatment against prostate antigens | Day 28 post vector injection
  Day 7,14,21 and 28 post vector injection
To assess changes in PSA levels as a surrogate marker for prostate cancer following Ad.hIL-12 gene therapy | 1 week after vector injection
  1,2,4,6 and 8 weeks after vector injection
To assess changes in PSA levels as a surrogate marker for prostate cancer following Ad.hIL-12 gene therapy | 2 weeks after vector injection
  1,2,4,6 and 8 weeks after vector injection
To assess changes in PSA levels as a surrogate marker for prostate cancer following Ad.hIL-12 gene therapy | 4 weeks after vector injection
  1,2,4,6 and 8 weeks after vector injection
To assess changes in PSA levels as a surrogate marker for prostate cancer following Ad.hIL-12 gene therapy | 6 weeks after vector injection
  1,2,4,6 and 8 weeks after vector injection
To assess changes in PSA levels as a surrogate marker for prostate cancer following Ad.hIL-12 gene therapy | 8 weeks after vector injection
  1,2,4,6 and 8 weeks after vector injection

CONTACTS AND LOCATIONS:
Overall Officials: Simon Hall, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai